CLINICAL TRIAL: NCT01772992
Title: CVCTPlus: A Couples-Based Approach to Linkage to Care and ARV Adherence
Acronym: CVCTPLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Emory University (Other)
Responsible Party: Principal Investigator, Robert Stephenson, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00065111; 1R01HD075655-01A1 (NIH)
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: HIV couples adherence linkage to care viral suppression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (iVCT) (No Intervention): Male couples randomized to the control group (iVCT) will each receive individual HIV counseling and testing, separately.These couples in the control group (iVCT) will return every 6 months, up to 18 months, for individual visits, in which they will have STI testing and repeat HIV testing. All follow-up visits will be conducted separately.
- Experimental group (CVCTPLUS) (Experimental): Male couples randomized to the experimental group (CVCTPLUS) will each receive HIV counseling and testing as a couple. These couple will return for two additional visits that members of the control arm do not get, for two one-hour sessions of the Partner-STEPS. Couples in the experimental group (CVCTPLUS) at 8 and 10 weeks after the initial enrollment. They will also return every 6 months, up to 18 months, for visits in which they will be seen as a couple, in which they will have STI testing and repeat HIV testing. All follow-up visits will be conducted for the couples together.
  Interventions: Behavioral: CVCTPLUS

INTERVENTIONS:
Behavioral: CVCTPLUS — For the intervention, couples will receive HIV testing and counseling together as a dyad, and some couples will receive ARV adherence counseling (Partner-STEPS) together as a dyad.
  Other Names: Dyadic STEPS; Partner STEPS
  Arms: Experimental group (CVCTPLUS)

SUMMARY:
Men who have sex with men (MSM) continue to be the most heavily-impacted risk group in the US HIV epidemic. Studies suggest that the majority of incident HIV infections among MSM are attributable to sex with a main male sex partner. However, HIV prevention interventions that target male-male couples are lacking. Because of this, Couples HIV Voluntary Counseling and Testing (CVCT), an intervention that has been repeatedly shown to reduce HIV transmission within heterosexual couples, has been adapted to US MSM couples. Additionally, novel evidence demonstrates that antiretroviral therapy (ART) not only reduces morbidity and mortality among HIV-positive persons, but also serves to reduce the risk of HIV transmission to a negative partner by 96%. As adherence to ART is modifiable and levels of peer support have been shown to increase ART adherence, this current study proposes to use CVCT combined with dyadic adherence counseling ("CVCTPlus") to improve linkage to care, retention in care, ART adherence, and viral suppression among male-male couples using a cohort of 350 serodiscordant (one HIV(+) partner, one HIV(-) partner) couples in the greater Atlanta, Chicago, and Boston areas. Prospective couples (175 in each arm) will be followed for 18 months. At each visit, they will receive HIV testing, and both partners will complete a study survey measuring social and behavioral factors that may influence adherence, such as a couple's coping ability and their concordance of agreements regarding outside sex partners. Additionally, couples in the intervention arm will receive two additional sessions of Partner-STEPS.

DETAILED DESCRIPTION:
Since the earliest reports of AIDS in the United States, men who have sex with men (MSM) have been, and continue to be, the most heavily impacted risk group in the US HIV epidemic. In 2009, MSM accounted for 61% of new HIV diagnoses, an increase from 53% of HIV incidence in 2006. The "test and treat" strategy for HIV infection entails universal testing with immediate treatment for those who test seropositive, with the aim of achieving viral suppression among positives. The efficacy of treatment as prevention demonstrated in HPTN 052 has reinvigorated the discussion over using a "test and treat" strategy to reduce the incidence of HIV infection in the US. However, engagement-in-care research raises a note of caution regarding potential pitfalls in the effectiveness of this strategy. The recently published MMWR "Vital Signs" Report, showed only 28% of all HIV-infected persons in the US has a suppressed viral load. The estimates published by Gardner show that of the estimated 1.1 million persons infected with HIV in the United States, 21% of HIV-infected persons are currently undiagnosed. Of those who are diagnosed, losses occur at initial linkage to care and later in care such that only 50% remain in care, such that only 19% of HIV-infected persons in the US currently having viral load below the limits of assay detection. There is now substantial evidence of the role of couples - or main partnerships - in fueling the HIV epidemic among MSM in the US. A recent CDC analysis found that 68% of new infections among MSM in the US were ascribed to main sex partners, and the proportion of new infections from main sex partners was even higher among younger MSM. Led by Sullivan and Stephenson, recent work has illustrated the feasibility of enrolling couples into HIV prevention efforts and demand for couples-focused services among MSM. A response to the growing demand for couples-focused services has been the adaptation of Couples Voluntary Counseling and Testing (CVCT) for MSM in the US. A recent NIMH-funded RCT of CVCT versus traditional VCT among MSM (Sullivan PI) showed 22% of MSM couples to be sero-discordant. This collective evidence provides the foundation for the proposed activities. We know that a significant proportion of new HIV infections occur within couples, and we know that current levels of linkage to care, retention in care and adherence to ARVs are below par among US MSM. In April 2012, WHO released new guidelines for Couples HIV testing and counseling, including ARV for treatment and prevention among sero-discordant couples [7]. The guidelines report a significant gap in evidence around the uptake and adherence to ARV among couples, and the role of CVCT in shaping uptake and adherence to ARVs: the proposed research has the potential to add significantly to our understanding of these issues. The proposed activities investigate the utility of CVCT combined with dyadic adherence counseling for improving linkage to care, retention in care and adherence to ARVs. Through the screening of 350 MSM couples and the enrollment of couples in a RCT, the study aims to examine the impact of CVCTPlus (CVCT plus dyadic adherence counseling) versus the current standard of care (individual testing only) on linkage to HIV care, retention in HIV care, adherence to ARV and achievement of viral suppression among sero-discordant MSM couples. The specific aims are:

Primary Aims:

1. i. Aim 1: Examine if testing together for HIV and receiving dyadic adherence counseling (Partner-STEPS) increases linkage to care as defined as: within three months after HIV diagnosis, having (1) at least one clinical care appointment, (2) at least one CD4 count test performed, and (3) at least one viral load test performed

ii. Aim 2: Examine if testing together for HIV and receiving dyadic adherence counseling (Partner-STEPS) increases retention in care, as defined as: within the past 12 months, having (1) at least two routine HIV care visits at least three months apart, (2) two or more CD4 tests, and (3) two or more viral load tests

iii. Aim 3: Examine if testing together for HIV and receiving dyadic adherence counseling (Partner-STEPS) increases adherence to anti-retroviral therapy and reductions in viral loads / achievement of viral suppression

iv. Aim 4: Examine if testing together for HIV decreases sexual risk-taking both within dyads and with outside sexual partners

v. Aim 5: Examine if testing together increases couples' coping and communication abilities

Hypothesis: Couples who receive a package of CVCT and a dyadic-focused adherence intervention will achieve greater linkage to care, retention in care, adherence to ARVs and viral suppression than couples who receive the standard of care (individualized VCT and adherence counseling).

With increasing evidence of the role of ARVs in reducing HIV transmission, MSM couples represent a significant target group for new interventions. The proposed activities will provide new information demonstrating the efficacy of using a couples-based approach for increasing ARV adherence and care seeking among couples.

ELIGIBILITY:
b. Inclusion Criteria i. Male sex at birth ii. Male gender iii. 18 or older iv. Living in Atlanta, Chicago, or Boston for at least three months v. Has a main Male Sexual Partner of relationship duration one month or longer vi. In a known or assumed serodiscordant relationship, that is, where one member of the couple is HIV-positive and one is either known to be or believed to be HIV-negative or of unknown HIV status vii. If HIV-positive, reporting of one or more of the following forms of suboptimal HIV medication adherence:

1. Never having seen a prescribing provider for HIV care
2. Not having a viral load test performed in the past six months, or not knowing if a viral load test has been performed in the past six months
3. Never having been prescribed anti-HIV medications
4. Never having begun taking anti-HIV medications
5. Adherence to 90% or less of anti-HIV medications in the past week viii. No recent (one-year) severe intimate partner violence reported within the couple (note: mutually agreed-upon BDSM practices are excluded and not analogous with experiences of IPV)

(1) In the past six months, has he: i. Punched, hit or slapped you? ii. Kicked you? iii. Pushed or shoved you? iv. Used force or threats of force to make you do something sexual that you didn't want to do? v. Raped you? ix. No coercion to test for HIV reported within the couple x. Willingness to be tested for HIV with one's male sexual partner xi. Willingness to be randomized to either study arm xii. Participant reports feeling safe in his relationship

c. Exclusion Criteria i. Sex at birth other than male ii. Gender other than male iii. Either partner aged 17 or younger iv. Either partner living outside the Atlanta, Chicago, or Boston areas, or having moved to these areas within the past three months v. Does not have a main male sex partner or has a main male sex partner of relationship duration less than one month vi. Both partners have known or assumed negative HIV status vii. Both partners have known or assumed positive HIV status viii. Either partner reports experiencing or perpetrating severe physical or sexual intimate partner violence within the couple within the past year (see above, note that consensual BDSM practices are not classified as IPV) ix. Either partner reports feeling unsafe in his relationship x. Either partner reports feeling coerced or pressured into testing for HIV xi. Either partner reports feeling coerced or pressured into joining the research study xii. Unwillingness to test for HIV together with one's sexual partner xiii. Unwillingness to be randomized

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Linkage to Care | 18 months
  within three months after HIV diagnosis, having (1) at least one clinical care appointment, (2) at least one CD4 count test performed, and (3) at least one viral load test performed

SECONDARY OUTCOMES:
Retention in care | 18 months
  within the past 12 months, having (1) at least two routine HIV care visits at least three months apart, (2) two or more CD4 tests, and (3) two or more viral load tests

OTHER OUTCOMES:
Viral suppression | 18 months
  For each study visit we will extract viral load and CD4 counts from the positive participant's medical record. If there are multiple reports within 30 days of the study visit, we will use the count nearest in date to the study visit. If there is no report within 30 days of the study visit, this will be treated as missing data. In the case of the sero-conversion of a negative partner, we will also collect viral load and CD4 counts from the newly positive partner at each study visit. Viral suppression will be considered achieved if the medical records report a viral load below the level of detection for the site specific assay
Decrease sexual risk-taking | 18 months
  At each follow-up visit, each partner will be asked about unprotected anal intercourse that occurs within the partnership during the previous follow-up period.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rollins School of Public Health, Emory University, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Harvard School of Public Health, Boston, Massachusetts
  - Fenway Health Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Stephenson R, Suarez NA, Garofalo R, Hidalgo MA, Hoehnle S, Thai J, Mimiaga MJ, Brown E, Bratcher A, Wimbly T, Sullivan P. Project Stronger Together: Protocol to Test a Dyadic Intervention to Improve Engagement in HIV Care Among Sero-Discordant Male Couples in Three US Cities. JMIR Res Protoc. 2017 Aug 31;6(8):e170. doi: 10.2196/resprot.7884. PMID 28860107